CLINICAL TRIAL: NCT00682630
Title: Phase I, Randomized, Single Dose, Bioequivalence Trial of Pyronaridine Artesunate To-be-marketed Tablet to the Clinical Trial Reference Tablet
Brief Title: Bioequivalence Trial of Pyronaridine Artesunate To-be-marketed Tablet to the Clinical Trial Reference Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-009-07
Record Dates: First submitted 2008-05-19; First posted 2008-05-22 (Estimated); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Malaria
Keywords: Malaria; anti-malarial; pyronaridine; pyronaridine artesunate (Pyramax); artemisinin based combination therapy (ACT)
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical Trial Reference Tablets first, then To-Be-Marketed Tablets (Experimental): Participants first received clinical trial reference 720:240 mg tablets on Day 0. After a washout period of 43 days, they then received to-be-marketed 720:240 mg tablets on Day 43, with a follow-up period of 42 days.
  Interventions: Drug: pyronaridine artesunate clinical trial reference tablets; Drug: pyronaridine artesunate to-be-marketed tablets
- To-Be-Marketed Tablets first, then Clinical Trial Reference Tablets (Experimental): Participants first received to-be-marketed 720:240 mg tablets on Day 0. After a washout period of 43 days, they then received clinical trial reference 720:240 mg tablets on Day 43, with a follow-up period of 42 days.
  Interventions: Drug: pyronaridine artesunate clinical trial reference tablets; Drug: pyronaridine artesunate to-be-marketed tablets

INTERVENTIONS:
Drug: pyronaridine artesunate clinical trial reference tablets — Single total oral dose of 720:240 mg (4 tablets of 180:60 mg)
  Other Names: Pyramax; PA
Drug: pyronaridine artesunate to-be-marketed tablets — Single total oral dose of 720:240 mg (4 tablets of 180:60 mg)
  Other Names: Pyramax; PA

SUMMARY:
The primary objective of this study is to determine the bioequivalence of the combination of pyronaridine and artesunate (180:60mg) to-be-marketed tablet to the clinical trial reference tablet administered as a single total dose of 720:240 mg in healthy adults. The secondary objective is to assess the safety of the two formulations.

DETAILED DESCRIPTION:
This is a phase I, randomized, single dose, two-way cross-over study of two tablet formulations of the combination of pyronaridine and artesunate (180:60 mg). The study will include 42 healthy participants, comprising male and female adults.

Participants will be randomized to receive either reference tablet formulation or to-be-marketed formulation first and then will be crossed over to receive the opposite Intervention. The study will consist of two single dose treatments of 720:240 mg tablets, separated by a washout period of 43 days.

Participants will go to the clinic the evening before dosing (dosing days were Day 0 for period 1 and Day 43 for period 2) under fasting condition and remain in the hospital for 24 hours after receiving dosing.

Participants will stay in the hospital for 24 hours after their arrival at the clinic. They will return to the clinic at Day 2, 3, 5, 7, 14, 21, 28, 35 and 42 on an ambulatory basis. At Day 43, the dosing for the second sequence will start and a similar schedule of visits will be followed. Each participant will be followed-up for an additional 42 days after the start of the second study period, until the final visit (Day 85). The total duration of participation is 85 days plus a maximum of 2 weeks screening period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18 and 45 years with a body weight between 55 and 75 kg and a body mass index using Quetelet's Index - weight (kg)/height2 (m2) between 18-28
2. Signed and dated written informed consent form before undergoing any study related activities, including discontinuation of any prohibited medications
3. Medically normal subjects with no significant abnormal findings at the screening physical examination as evaluated by the clinical investigator
4. Normal (or abnormal and clinically insignificant) laboratory values at screening
5. Female subjects of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who was post-menopausal (i.e., one year without menses)
6. Female subjects of childbearing potential with a negative urine pregnancy test at screening and who agreed to one of the accepted forms of contraception
7. The ability to understand the requirements of the study and willingness to comply with all study procedures

Exclusion Criteria:

1. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, acute QTc interval greater or equal to 450 mseconds), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other abnormality (including head trauma)
2. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine or artesunate or other artemisinins
3. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
4. Known seropositive HIV antibody
5. Previous participation in any clinical trial with pyronaridine artesunate
6. Presence or recent history (last two years) of tobacco abuse (≥10 cigarettes/day)
7. Known or suspected alcohol abuse or illicit drug use 10 years before the study start or positive findings on urine drug screen
8. Intake of alcoholic beverages or caffeine-containing food or beverages, such as coffee, tea, chocolate, or cola, 24 h before study drug administration
9. Use of over-the-counter (OTC) medications, including vitamins, analgesics, or antacids, 72 h before the study start
10. Use of prescription medications 14 days before the study start or required chronic use of any prescription medication
11. Use of enzyme-altering agents (e.g., barbiturates, phenothiazines, cimetidine, etc.) 30 days before the study start
12. Plasma donation 3 months before the study start
13. Blood donation of 500 mL or more 3 months before the study start
14. Participation in an investigational drug study 3 months before randomization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Borghini Fuhrer, PhD, Study Director — Medicines for Malaria Venture
Locations (1):
- Cross Research S.A., Phase I Unit, Arzo, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (Day 0)
Arm/Group | Clinical Trial Reference Tablets First, Then To-Be-Marketed Tablets | To-Be-Marketed Tablets First, Then Clinical Trial Reference Tablets
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Period: Washout (43 Days)
Arm/Group | Clinical Trial Reference Tablets First, Then To-Be-Marketed Tablets | To-Be-Marketed Tablets First, Then Clinical Trial Reference Tablets
Started | 20 | 21
Completed | 18 | 19
Not Completed | 2 | 2
Period: Second Intervention (Day 43)
Arm/Group | Clinical Trial Reference Tablets First, Then To-Be-Marketed Tablets | To-Be-Marketed Tablets First, Then Clinical Trial Reference Tablets
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: Follow-up (42 Days)
Arm/Group | Clinical Trial Reference Tablets First, Then To-Be-Marketed Tablets | To-Be-Marketed Tablets First, Then Clinical Trial Reference Tablets
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all subjects who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Trial Reference Tablets First, Then To-Be-Marketed Tablets | To-Be-Marketed Tablets First, Then Clinical Trial Reference Tablets | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (7.8) | 33.5 (4.9) | 33.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.5 (1.4) | 23.3 (3.0) | 23.4 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Pyronaridine Pharmacokinetics: Tmax, Half-life
Description: Tmax: time to maximum concentration Half-life: computed as ln (2)/kel
Time Frame: Sampling performed at predose at 0 h and at, 0.5, 1, 1.5, 2.5, 4, 6, 8, 12, 24, 48, 72 h and on Day 5, 7, 14, 21, 28, 35, 42 for each period
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: days
Groups:
- Clinical Trial Reference Tablets: Participants who received clinical trial reference 720:240 mg tablets in either state each morning in either the first intervention (Day 0) or the second intervention (Day 43).
- To-Be-Marketed Tablets: Participants who received to-be-marketed 720:240 mg tablets in either state each morning in either the first intervention (Day 0) or the second intervention (Day 43).
Arm/Group | Clinical Trial Reference Tablets | To-Be-Marketed Tablets
Number analyzed (Participants) | 40 | 39
days
  Tmax | 0.184 (0.145) | 0.166 (0.131)
  Half-life | 14.2 (5.28) | 14.1 (4.00)

2. Primary Outcome: Pyronaridine (PP), Artesunate (AS), Dihydroartemisinin (DHA) Pharmacokinetics: Cmax
Description: Cmax: maximum peak observed concentration
Time Frame: PP sampling performed at predose at at 0 h and at, 0.5, 1, 1.5, 2.5, 4, 6, 8, 12, 24, 48, 72 h and on Day 5, 7, 14, 21, 28, 35, 42 for each period AS, DHA sampling performed at predose at 0 h and at 0.25, 0.5, 1, 1.5, 2.5, 4, 6, 8, 12 h for each period
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Clinical Trial Reference Tablets | To-Be-Marketed Tablets
Number analyzed (Participants) | 40 | 39
ng/ml
  PP Cmax | 512 (183) | 533 (190)
  AS Cmax | 183 (175) | 154 (101)
  DHA Cmax | 987 (476) | 959 (356)

3. Primary Outcome: Artesunate (AS) and Dihydroartemisinin (DHA) Pharmacokinetics: Tmax, Half-life
Description: Tmax: time to maximum concentration Half-life: computed as ln (2)/kel
Time Frame: Sampling performed at predose at 0 h and at 0.25, 0.5, 1, 1.5, 2.5, 4, 6, 8, 12 h for each period
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Clinical Trial Reference Tablets | To-Be-Marketed Tablets
Number analyzed (Participants) | 40 | 39
hours
  AS Tmax | 0.488 (0.226) | 0.548 (0.279)
  DHA Tmax | 1.14 (0.555) | 1.39 (0.823)
  AS half-life | 0.549 (0.447) | 0.538 (0.717)
  DHA half-life | 1.53 (0.452) | 1.84 (0.571)

4. Primary Outcome: Pyronaridine Pharmacokinetics: AUC0-last, AUC0-∞
Description: AUC0-last: Area under the concentration-time curve from time 0 (0 h) through the last quantifiable concentration time (LQCT), where LQCT is the time at which the last sample with a quantifiable concentration was drawn AUC0-∞: Area under the concentration-time curve from time 0 (0 h) to infinity, computed using the linear trapezoidal rule as AUClast + CLQCT / Kel
Time Frame: as for outcome 1
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng*day/ml
Arm/Group | Clinical Trial Reference Tablets | To-Be-Marketed Tablets
Number analyzed (Participants) | 40 | 39
ng*day/ml
  AUC0-last | 729 (216) | 762 (272)
  AUC0-∞ | 877 (244) | 904 (291)

5. Primary Outcome: Artesunate (AS) and Dihydroartemisinin (DHA): AUC0-last, AUC0-∞
Description: as for outcome 4
Time Frame: Sampling performed at predose at 0 h and at 0.25, 0.5, 1, 1.5, 2.5, 4, 6, 8, 12 h for each period
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Clinical Trial Reference Tablets | To-Be-Marketed Tablets
Number analyzed (Participants) | 40 | 39
ng*hr/ml
  AS AUC0-last | 139 (106) | 121 (79.7)
  DHA AUC0-last | 2150 (889) | 2120 (834)
  AS AUC0-∞ | 155 (107) | 137 (83.9)
  DHA AUC0-∞9 | 2166 (896) | 2143 (849)

ADVERSE EVENTS:
Time Frame: 85 days (43 days Period 1, 42 days Period 2)
Description: AE reporting was assessed through direct questioning.
Arm/Group | To-Be-Marketed Tablets | Clinical Trial Reference Tablets
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 26/39 | 28/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | To-Be-Marketed Tablets (N=39) | Clinical Trial Reference Tablets (N=40)
Abdominal discomfort (Gastrointestinal disorders) | 9 (9) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (14) | 15 (15)
Vomiting (Gastrointestinal disorders) | 15 (17) | 12 (15)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 8 (8)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No